CLINICAL TRIAL: NCT02237274
Title: Cardiopulmonary Adaptation of Short Term Exposure to High Altitude in Fontan Patients: Swiss Fontan & ALtitude COllaboratioN (FALCON) Study
Acronym: FALCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Mach Gaensslen Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 222/13
Record Dates: First submitted 2014-08-26; First posted 2014-09-11 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Fontan Procedure; Altitude
Keywords: Fontan circulation; High altitude exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with Fontan circulation (Experimental): High altitude exposition
  Interventions: Other: High altitude exposition
- Age and gender-matched healthy volunteers (Other): High altitude exposition
  Interventions: Other: High altitude exposition

INTERVENTIONS:
Other: High altitude exposition — High altitude exposition

SUMMARY:
Important advances in cardiac surgery, intensive care, and diagnostic modalities over the last decades have led to a steady growth in the number of adults with congenital heart defects. Among adults with congenital heart disease, patients with a Fontan circulation typically show the lowest values of peak oxygen consumption. For these patients, strict exclusion from activities at high altitude may have an impact on quality of life. The investigators aim to elucidate the short term effects of a stay at high altitude on hemodynamic adaptation, exercise capacity and clinical well being in adult Fontan patients. The investigators hypothesize that patients with a Fontan circulation in NYHA functional class I-II are able to increase their cardiac output during exercise at high altitude in order to meet the required metabolic demands and therefore tolerate the journey to the Jungfraujoch well.

DETAILED DESCRIPTION:
Background:

Important advances in cardiac surgery, intensive care, and diagnostic modalities over the last decades have led to a steady growth in the number of adults with congenital heart defects (Grown-up congenital heart disease GUCH). Among adults with congenital heart disease, patients with a Fontan circulation typically show the lowest values of peak oxygen consumption with peak VO2 values between 15 and 29 ml/kg/min, corresponding to 43-64 % of the predicted values in healthy controls. For these patients, strict exclusion from activities at high altitude may have an impact on quality of life. Unfortunately, the most recent recommendations for physical activity, recreation sport, and exercise training in paediatric patients with congenital heart disease do not provide specific recommendations. The investigators study therefore aims to elucidate the short term effects of a stay at high altitude on hemodynamic adaptation, exercise capacity and clinical well being in adult Fontan patients. These results are necessary to counsel GUCH patients with respect to their leasure activities in Switzerland.

Objective:

The aims of the study are to measure a)the hemodynamic adaptation (pulmonary blood flow) at rest and during exercise; b)the response of cardiopulmonary parameters to exercise (ventilation, O2 uptake) and c) heart rate variability and occurrence of arrhythmias during the journey and while performing study measures in patients with a Fontan circulation. The measurements will be performed at high altitude and at lowland and compared with an age- and gender-matched control group of healthy subjects. The objective is to test the clinical tolerance of high altitude exposure after a rapid ascent with public transport in patients with a Fontan circulation. The investigators hypothesize that patients with a Fontan circulation in NYHA functional class I-II are able to increase their cardiac output during exercise at high altitude in order to meet the required metabolic demands despite hypoxia induced pulmonary vasoconstriction and therefore tolerate the journey to the Jungfraujoch well.

Methods:

The investigators aim to include 30 patients with a Fontan circulation and 30 age and gender-matched healthy adults. Baseline testing in Bern (540m over sea level)includes: a symptom limited cardiopulmonary exercise stress test on a cycle ergometer with a ramp protocol (CPX); a pulmonary function test (spirometry); a symptom limited, stepwise increasing workload test with non-invasive inert gas rebreathing method for pulmonary blood flow measurement during exercise (Innocor®); analysis of heart rate variability (HRV); Holter-ECG monitoring for detection of arrhythmias.

Within a time period of 12 weeks, the baseline tests will be repeated on the Jungfraujoch (3454m).

The primary endpoint of this study is the increase of pulmonary blood flow during exercise in response to high altitude exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18years
* Congenital heart disease and Fontan circulation
* NYHA functional class I & II
* Peak VO2 > 45% of predicted
* Signed informed consent

Exclusion Criteria:

* "Failing Fontan", peak VO2 < 45% of predicted
* Significant right-to-left shunt
* Baseline arterial O2 saturation at rest <90% at room air
* Hospitalization within the last 3 months for cardiac reasons
* Decrease in functional NYHA class within the last 3 months
* Motor skill inability to perform a maximal exercise stress test
* Respiratory Exchange Ratio < 1
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pulmonary blood flow during exercise at high altitude | During exercise at high altitude, maximum 12 weeks after baseline measurements
  Pulmonary blood flow measurement during exercise: a symptom limited, stepwise increasing workload test with non-invasive inert gas rebreathing method for (Innocor®)

SECONDARY OUTCOMES:
Change from baseline in peak VO2 (exercise capacity) | During exercise at high altitude, maximum 12 weeks after baseline measurements
  Peak VO2 (exercise capacity): a symptom limited cardiopulmonary exercise stress test on a cycle ergometer with a ramp protocol (CPX)
Change from baseline in clinical symptoms (tolerance of high alt. exposure, funct.l NYHA class, dyspnea Borg scale) | During exercise at high altitude, maximum 12 weeks after baseline measurements
Change from baseline in sympathovagal balance of the autonomic nervous system | During exercise at high altitude, maximum 12 weeks after baseline measurements
Change from baseline in occurrence of arrhythmias | During exercise at high altitude, maximum 12 weeks after baseline measurements
  Measured by holter-ECG monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schwerzmann, Professor, Dr med., Principal Investigator — Department of Cardiology, GUCH, Bern University Hospital
Locations (1):
- Department of Cardiology, GUCH, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Result] Bartsch P, Gibbs JS. Effect of altitude on the heart and the lungs. Circulation. 2007 Nov 6;116(19):2191-202. doi: 10.1161/CIRCULATIONAHA.106.650796. No abstract available. PMID 17984389
- [Result] Fredriksen PM, Veldtman G, Hechter S, Therrien J, Chen A, Warsi MA, Freeman M, Liu P, Siu S, Thaulow E, Webb G. Aerobic capacity in adults with various congenital heart diseases. Am J Cardiol. 2001 Feb 1;87(3):310-4. doi: 10.1016/s0002-9149(00)01364-3. PMID 11165966
- [Result] Driscoll DJ, Durongpisitkul K. Exercise testing after the Fontan operation. Pediatr Cardiol. 1999 Jan-Feb;20(1):57-9; discussion 60. doi: 10.1007/s002469900397. No abstract available. PMID 9861079
- [Result] Freedom RM, Hamilton R, Yoo SJ, Mikailian H, Benson L, McCrindle B, Justino H, Williams WG. The Fontan procedure: analysis of cohorts and late complications. Cardiol Young. 2000 Oct;10(4):307-31. doi: 10.1017/s1047951100009616. No abstract available. PMID 10950328
- [Result] Takken T, Giardini A, Reybrouck T, Gewillig M, Hovels-Gurich HH, Longmuir PE, McCrindle BW, Paridon SM, Hager A. Recommendations for physical activity, recreation sport, and exercise training in paediatric patients with congenital heart disease: a report from the Exercise, Basic & Translational Research Section of the European Association of Cardiovascular Prevention and Rehabilitation, the European Congenital Heart and Lung Exercise Group, and the Association for European Paediatric Cardiology. Eur J Prev Cardiol. 2012 Oct;19(5):1034-65. doi: 10.1177/1741826711420000. PMID 23126001
- [Result] Rimoldi SF, Sartori C, Seiler C, Delacretaz E, Mattle HP, Scherrer U, Allemann Y. High-altitude exposure in patients with cardiovascular disease: risk assessment and practical recommendations. Prog Cardiovasc Dis. 2010 May-Jun;52(6):512-24. doi: 10.1016/j.pcad.2010.03.005. PMID 20417345
- [Result] Luks AM, Stout K, Swenson ER. Evaluating the safety of high-altitude travel in patients with adult congenital heart disease. Congenit Heart Dis. 2010 May-Jun;5(3):220-32. doi: 10.1111/j.1747-0803.2010.00415.x. PMID 20576041
- [Derived] Staempfli R, Schmid JP, Schenker S, Eser P, Trachsel LD, Deluigi C, Wustmann K, Thomet C, Greutmann M, Tobler D, Stambach D, Wilhelm M, Schwerzmann M. Cardiopulmonary adaptation to short-term high altitude exposure in adult Fontan patients. Heart. 2016 Aug 15;102(16):1296-301. doi: 10.1136/heartjnl-2016-309682. Epub 2016 May 23. PMID 27217067